CLINICAL TRIAL: NCT04424849
Title: Initial Thoracic CT Findings and Mechanical Ventilation Requirement in Patients Admitted to Intensive Care Unit With COVID-19
Brief Title: Thorax Computed Tomography Severity Score and Outcome in COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kazim Rollas, MD, Tepecik Training and Research Hospital
Other Study IDs: 2020/5-4
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients: Patient tested positive for COVID-19 who had a CT scan
  Interventions: Diagnostic Test: CT-Scan

INTERVENTIONS:
Diagnostic Test: CT-Scan — Chest CT scan on admission to the intensive care unit

SUMMARY:
The most common thorax Computed tomography (CT) findings are multifocal ground-glass opacities and peripheral consolidation in patients with COVID-19. Septal thickening, bronchiectasis, pleural thickening, and subpleural involvement may also be observed. Although these findings are not specific to COVID-19, the severity of pulmonary involvement is expected to be correlated with thorax CT findings.

DETAILED DESCRIPTION:
Thorax computed tomography severity score defined by Yang et al. can be used to evaluate the severity of pulmonary involvement in COVID-19 patients. We aimed to investigate whether the initial thorax computed tomography severity score can predict mechanical ventilation requirement and mortality in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* COVID-19 confirmed by positive RT-PCR and/or antibody testing
* CT scan at intensive care unit admission

Exclusion Criteria:

* Loss of CT data
* Chronic lung disease findings by CT that may lead to misinterpretation
* RT-PCR results unavailable or negative
* Terminal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to the intensive care unit with COVID-19 pneumonia confirmed by RT-PCR
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Invasive respiratory support in patients with COVID-19 | 120 days
  Whether Thorax CT findings predict invasive mechanical ventilation requirement of covid-19 patients

SECONDARY OUTCOMES:
Mortality in patients with COVID-19 | 120 days
  Whether Thorax CT findings predict mortality of covid-19 patients

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No